CLINICAL TRIAL: NCT05415514
Title: Feasibility Study of the Instrumented Evaluation of Eccentric Strengthening in Paresis Patients
Acronym: RE PAR EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC22_0173
Record Dates: First submitted 2022-06-07; First posted 2022-06-13 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Paralysis
MeSH Terms: conditions — Paralysis

STUDY DESIGN:
Intervention Model Description: instrumented evaluations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Instrumented assessment of muscle function (Other): During the instrumented evaluations, the investigators will evaluate the possibility of measuring the passive and active function of the muscle using: - an isokinetic dynamometer, an ultrasound and elastography device, an electrical stimulation of the calf nerve
  Interventions: Other: Instrumented assessment of muscle function

INTERVENTIONS:
Other: Instrumented assessment of muscle function — During the instrumented evaluations, we will evaluate the possibility of measuring the passive and active function of the muscle using: - an isokinetic dynamometer, an ultrasound and elastography device, an electrical stimulation of the calf nerve

SUMMARY:
he aim of the "RE PAR EX" research is to evaluate the feasibility of the instrumented examination of the effects of eccentric muscle strengthening in paralytic patients. This project is part of the research axis of the movement analysis laboratory.

Following a stroke or spinal cord injury, patients develop a spastic paresis syndrome, which is characterized by the appearance of paresis, musculo-tendinous retractions and muscular hyperactivities.

If the traditional treatments proposed (stretching, motor work) show limits, the use of eccentric muscle strengthening in paresis patients has been developing for about ten years, with results superior to the usual treatments. The results of the studies evaluating it are focused on clinical evaluations and do not make it possible to identify the precise origin of the observed responses.

A pathophysiological understanding of the therapeutic effects of eccentric strengthening would be possible through instrumented examination of muscle structure and function, combining dynamometry, ultrasound, elastrography and electromyography (EMG). However, the feasibility of this quantified instrumental examination in paretic patients during a strengthening protocol has not been evaluated.

The feasibility of a quantified instrumented examination in this setting is the aim of this research, a necessary prerequisite for a larger interventional study to evaluate the biomechanical and neurophysiological effects of eccentric muscle strengthening in paretic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 80 years;
* Validation by the medical team of an eccentric strengthening protocol:

presence of a paresis of the studied muscle considered as functionally (triceps surae rated at 2 or more on the MRC scale), more or less associated with HAM and muscl retraction;

* Patient with a traumatic or ischemic spinal cord injury of grade Asia Impairment Scale (AIS) C or D (incomplete motor impairment) < 6 months or stroke < 6 months;
* Patient is competent to consent (Boston Diagnostic Aphasia Examination [BDAE] score greater than or equal to 2);
* Patient hospitalized in the neurological PRM service of the Nantes University Hospital.

Exclusion Criteria:

* History of functional surgery < 3 months ;
* Patient with osteoarticular lesions considered as a contraindication to to rehabilitation;
* Patient who is unlikely to adhere to the study program and/or not compliant compliant in the judgment of the investigator or refusing to participate in the study;
* Patients with a progressive pathology that contraindicates major muscular efforts (syrinx, cancer, etc.) (syrinx, cancer, cardiovascular instability...);
* Patients who are minors, protected adults, adults unable to express their consent or pregnant woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
proportion of usable data collected (ultrasound and elastographic images, EMG, force curves, etc.) compared to the expected usable data | 14 weeks

SECONDARY OUTCOMES:
To measure the duration of the examinations | 14 weeks
the average length of stay of included patients | 14 weeks
the patient's opinion through a self-questionnaire of satisfaction | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lecharte, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France